CLINICAL TRIAL: NCT06692192
Title: Role of Experience, Conscious Awareness, and Plasticity in Psilocybin's Behavioral Effects - Follow-Up Study (The RECAP 2 Study)
Brief Title: The RECAP2 Study: Midazolam and Psilocybin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Vail Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-0852; A538900 (Other: UW- Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW- Madison); Protocol Version 12/12/2025 (Other: UW- Madison)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Psilocybin
Keywords: sub-optimal wellbeing
MeSH Terms: interventions — Psilocybin; Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Psilocybin and intravenous (IV) midazolam (Experimental): Psilocybin (25 mg) + IV midazolam
  Interventions: Drug: Psilocybin; Drug: Midazolam
- Group 2: Psilocybin and IV saline (Experimental): Psilocybin (25 mg) + IV saline (placebo for midazolam)
  Interventions: Drug: Psilocybin; Drug: Saline
- Group 3: Psilocybin and IV midazolam (Experimental): Psilocybin (1 mg/control) + IV midazolam
  Interventions: Drug: Psilocybin; Drug: Midazolam
- Group 4: Psilocybin and IV saline (Experimental): Psilocybin (1 mg/control) + IV saline
  Interventions: Drug: Psilocybin; Drug: Saline

INTERVENTIONS:
Drug: Psilocybin — 25mg of psilocybin
  Other Names: Psilocybine; Psilocibin
  Arms: Group 1: Psilocybin and intravenous (IV) midazolam; Group 2: Psilocybin and IV saline
Drug: Psilocybin — 1mg of psilocybin
  Other Names: Psilocybine; Psilocibin
  Arms: Group 3: Psilocybin and IV midazolam; Group 4: Psilocybin and IV saline
Drug: Midazolam — The goal of the midazolam dosing regimen is to induce amnesia of the psychedelic experience without inducing over-sedation during the dosing session.
  Arms: Group 1: Psilocybin and intravenous (IV) midazolam; Group 3: Psilocybin and IV midazolam
Drug: Saline — Saline will be administered as a placebo for midazolam
  Arms: Group 2: Psilocybin and IV saline; Group 4: Psilocybin and IV saline

SUMMARY:
The goal of this clinical trial is to learn about the role that inducing neuroplasticity (the brain's ability to adapt and change) plays in the behavioral effects of psilocybin in people who have experienced a mild decline in emotional wellbeing.

Researchers will compare different doses of psilocybin combined with midazolam or placebo to see what dose induces increased wellbeing.

Participants will:

* Receive one of four possible combinations of medications
* Undergo an MRI
* Complete questionnaires
* Undergo transcranial magnetic stimulation (TMS) and EEG

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role that inducing neuroplasticity plays in the behavioral effects of psilocybin in people with modest decrements in emotional wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years at screening, of any identified gender and racial/ethnic group
* Physically healthy; does not meet criteria for an exclusionary medical condition
* English-speaking (able to provide consent and complete questionnaires)
* Modest decrement in self-reported wellbeing without the presence of a DSM-5 Axis I mood or anxiety disorder
* Able to undergo magnetic resonance imaging (MRI) and transcranial magnetic stimulation (TMS)

Exclusion Criteria:

* Exclusionary DSM-5 psychiatric diagnosis and/or active suicidal ideation
* Exclusionary medical conditions
* Clinically significant safety lab abnormalities (i.e., Complete Blood Count with Differential, Comprehensive Metabolic Panel, and urinalysis)
* Clinically significant electrocardiogram (ECG)
* Use of psychotropic or CNS-altering medications within 3 months of screening
* Hypertension or tachycardia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Warwick-Edinburgh Mental wellbeing Scale (WEMWBS) | Baseline to 7 days post-dose
  WEMWBS is a 14-item questionnaire in which participants describe their experience of each item. It is scored on a 5-point Likert scale, possible range of 14-70 where higher scores indicate higher levels of wellbeing.
Change in Brief Experiential Avoidance Questionnaire (BEAQ) | Baseline to 7 days post-dose
  The BEAQ is a 15-item questionnaire assessing participants agreement with wellbeing statements. It is scored on a 6-point Likert scale, ranging from 15-90 with higher scores indicating a greater tendency towards experiential avoidance
Change in Probabilistic Reversal Learning (PRL) | Baseline to 7 days post-dose
  Participants are presented with two stimuli or options and learn which one is more likely to be associated with a reward based on feedback after each trial. After a certain number of trials, the reward contingencies are reversed, meaning the previously advantageous option becomes less likely to be rewarded, and vice versa. The task assesses how quickly and effectively individuals can adapt to these changes in reward contingencies. Researchers analyze various performance metrics, such as the speed of reversal, the number of errors, and the patterns of choices (e.g., win-stay, lose-shift).
Change in transcranial magnetic stimulation evoked potential (TEP) amplitude | Baseline to 7 days post-dose
  TEP measures neural excitability in the stimulated region of the brain.

SECONDARY OUTCOMES:
Change in WEMWBS | Baseline to 28 days post-dose
  WEMWBS is a 14-item questionnaire in which participants describe their experience of each item. It is scored on a 5-point Likert scale, possible range of 14-70 where higher scores indicate higher levels of wellbeing.
Change in BEAQ | Baseline to 28 days post-dose
  The BEAQ is a 15-item questionnaire assessing participants agreement with wellbeing statements. It is scored on a 6-point Likert scale, ranging from 15-90 with higher scores indicating a greater tendency towards experiential avoidance
Change in PRL | Baseline to 28 days post-dose
  Participants are presented with two stimuli or options and learn which one is more likely to be associated with a reward based on feedback after each trial. After a certain number of trials, the reward contingencies are reversed, meaning the previously advantageous option becomes less likely to be rewarded, and vice versa. The task assesses how quickly and effectively individuals can adapt to these changes in reward contingencies. Researchers analyze various performance metrics, such as the speed of reversal, the number of errors, and the patterns of choices (e.g., win-stay, lose-shift).
Change in TEP amplitude | Baseline to 28 days post-dose
  TEP measures neural excitability in the stimulated region of the brain.
Altered States of Consciousness (ASC) questionnaire | Dosing 1 day
  Participants will complete a selection of several questions from the ASC questionnaire that strongly associate positively or negatively with later antidepressant effect of psilocybin in patients with treatment resistant depression or capture classic features of the psychedelic experience. During the dosing session, investigator will repeatedly ask selected items from the ASC scale to get a "real time" measure of what the participants are experiencing. Each of these items will be scored separately. Higher score are indicative of a more intense psychedelic experience.
Emotional Breakthrough Inventory (EBI) | Dosing 1 day
  The EBI is a 6-item scale that assesses the presence and severity of emotionally challenging/distressing experiences that occur during a psychedelic experience. Participants rate to what extent the statements apply to their experience by marking a single line across each scale. Scale ranges from not at all to very much so. Higher scores (more slashes toward the 'very much so' end) on the scale have been associated with enhanced well-being following psychedelic use
Psychological Insight Questionnaire (PIQ) | Dosing 1 day
  The PIQ is a 23-item instrument designed to query self-perceived attainment of insight during a psychedelic medicine session. Items are rated on a 6-point Likert scale, 0 = no not at all and 5 = extremely. Possible scares range from 0-115, with higher scores indicating greater insight.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No